CLINICAL TRIAL: NCT06317623
Title: Urinary Tract Dilations in Prenatal and Postnatal Life
Status: Recruiting | Type: Observational
Sponsor: SonoClinic (Network)
Responsible Party: Sponsor
Other Study IDs: 0292/21/2023-00590
Record Dates: First submitted 2024-02-26; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Urinary Tract Dilatation
Keywords: prenatal diagnosis; prenatal ultrasound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- UTD A1, low risk group: A group of fetuses and children with less severe dilation of the urinary tract in second or third trimester of pregnancy
  Interventions: Diagnostic Test: Prenatal and postnatal ultrasound examination
- UTD A2-3, high risk group: A group of fetuses and children with severe dilation of the urinary tract in second or third trimester of pregnancy
  Interventions: Diagnostic Test: Prenatal and postnatal ultrasound examination

INTERVENTIONS:
Diagnostic Test: Prenatal and postnatal ultrasound examination — Prenatal ultrasound examination of fetus with urinary tract dilation in second trimester and next in third trimester and when the dilation is persist, the child is managed after birth by pediatric nephrologist.

SUMMARY:
The goals of this study are to use a questionnaire survey to determine the state of awareness of the diagnosis and management of patients with urinary tract dilation across several medical professionals, to predict the severity of the postnatal course and surgical intervention in fetuses with urinary tract dilation detected during pregnancy, and to create a model of prenatal and postnatal care for patients with dilation of the urinary tract for multidisciplinary use.

DETAILED DESCRIPTION:
Currently, in Slovakia, a multidisciplinary standard of health care for patients with dilation of the urinary tract is not present. Prenatal diagnosis of anomalies of the urinary system includes the entire spectrum of anomalies, genetic diseases or anatomical deviations, which have a non-uniform classification and different terminology in a wide range of literature. Therefore, prenatal diagnosis of these anomalies, as well as dilation diseases of the urinary tract, in different centers is different, often subjective and outdated. However, some findings on the urinary tract, even with regard to the sex of the fetus, require great attention, defining the degree of severity and precisely targeted management, the task of which is to prevent serious complications in postnatal life. Dilative diseases of the urinary tract may not be clinically obvious after birth, but in the long term, if they are not detected, serious and irreversible kidney damage may occur. The goals of this study are therefore 1. to confuse the current situation in the multidisciplinary medical sector regarding the issue of dilations of the urinary tract; 2. in the conducted study to identify fetuses with such a degree of dilation of the urinary tract (according to the UTD classification from 2014) that requires stricter management in the prenatal and postnatal period and which are at high risk of surgical intervention postnatally and 3. subsequently create a model of health care for multidisciplinary cooperation for a patient with dilation of the urinary tract.

ELIGIBILITY:
Inclusion criteria:

* Singleton pregnant women whose fetuses were diagnosed with dilation of the urinary tract as an isolated US finding before the 28th week of pregnancy. Fetal patients with subsequent US control in the third trimester after the 28th week of pregnancy.
* Newborns and children with prenatally diagnosed UTD, which, depending on the severity, required a postnatal examination by a pediatric nephrologist within a month after birth and then in his follow-up up to 6 months after birth.

Exclusion criteria:

* Multiple pregnancies
* Urinary tract dilation in fetuses diagnosed in the third trimester
* Associated anomalies in fetuses
* Aneuploidy
* Newborns and children monitored by someone other than a selected pediatric nephrologist Patients who were lost from follow-up

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — fertility period of women
Study Population: Singleton pregnant women whose fetuses were diagnosed with dilatation of the urinary tract as an isolated finding before the 28th week of pregnancy. Dilatation of the urinary tract was categorized according to the 2014 UTD classification system.
  Newborns and children with prenatally diagnosed UTD, which, depending on the severity, required a postnatal check-up by a pediatric nephrologist within a month after birth and then in his follow-up up to 6 months after birth.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
The goal is the prediction of severe postnatal course and surgical intervention in fetuses with dilatation of the urinary tract according to the UTD classification created in 2014. | 20th week of pregnancy, 32th week of pregnancy, 2 days after birth, 6 months of child ´s life
  First part - Ultrasound examination of the fetus in the second trimester of pregnancy between the 18th and 24th weeks of pregnancy, no later than the 28th week of pregnancy.
  Examiner will be measure by ultrasound anteroposterior diameter renal pelvis in milimeters (mm).
  The second part - Classification of dilation of the urinary tract. The laterality and the detected finding is assigned the corresponding risk - for UTD A1 low risk, for UTD A2-3 high risk.
  Third part - Ultrasound control in the third trimester after the 32nd week of pregnancy. Renal pelvis will be examine by ultrasound and anteroposterior diameter will by measure in milimeters (mm).
  The fourth part - management of a child with UTD by a pediatric nephrologist. The child is followed in the study until the age of 6 months. Nephrologist will be measure anteroposterior diameter renal pelvis in milimeters (mm).

CONTACTS AND LOCATIONS:
Overall Officials: Svetlana Jánošová, Study Director — SonoClinic
Locations (1):
- Svetlana Jánošová, Záborské, Slovakia

IPD SHARING:
Plan to Share IPD: Yes
Data from ultrasound examination of fetusus will be share with other specialist from pediatric nephrology
Supporting Information: Study Protocol, CSR
Time Frame: After examination of fetuses in second trimester of pregnancy and 6 months after birth of child

REFERENCES:
- [Background] Nguyen HT, Herndon CD, Cooper C, Gatti J, Kirsch A, Kokorowski P, Lee R, Perez-Brayfield M, Metcalfe P, Yerkes E, Cendron M, Campbell JB. The Society for Fetal Urology consensus statement on the evaluation and management of antenatal hydronephrosis. J Pediatr Urol. 2010 Jun;6(3):212-31. doi: 10.1016/j.jpurol.2010.02.205. Epub 2010 Apr 15. PMID 20399145
- [Background] Nguyen HT, Benson CB, Bromley B, Campbell JB, Chow J, Coleman B, Cooper C, Crino J, Darge K, Herndon CD, Odibo AO, Somers MJ, Stein DR. Multidisciplinary consensus on the classification of prenatal and postnatal urinary tract dilation (UTD classification system). J Pediatr Urol. 2014 Dec;10(6):982-98. doi: 10.1016/j.jpurol.2014.10.002. Epub 2014 Nov 15. PMID 25435247
- [Background] Nguyen HT, Phelps A, Coley B, Darge K, Rhee A, Chow JS. 2021 update on the urinary tract dilation (UTD) classification system: clarifications, review of the literature, and practical suggestions. Pediatr Radiol. 2022 Apr;52(4):740-751. doi: 10.1007/s00247-021-05263-w. Epub 2022 Jan 4. PMID 34981177
- [Background] Mileto A, Itani M, Katz DS, Siebert JR, Dighe MK, Dubinsky TJ, Moshiri M. Fetal Urinary Tract Anomalies: Review of Pathophysiology, Imaging, and Management. AJR Am J Roentgenol. 2018 May;210(5):1010-1021. doi: 10.2214/AJR.17.18371. Epub 2018 Feb 15. PMID 29446682
- [Background] Sugar E, Gall J. [Orbital phlebography (author's transl)]. Fortschr Geb Rontgenstr Nuklearmed. 1974 Jul;121(1):20-4. No abstract available. German. PMID 4369632
- [Background] Braga LH, McGrath M, Farrokhyar F, Jegatheeswaran K, Lorenzo AJ. Society for Fetal Urology Classification vs Urinary Tract Dilation Grading System for Prognostication in Prenatal Hydronephrosis: A Time to Resolution Analysis. J Urol. 2018 Jun;199(6):1615-1621. doi: 10.1016/j.juro.2017.11.077. Epub 2017 Dec 2. PMID 29198999
- [Background] Nelson CP, Lee RS, Trout AT, Servaes S, Kraft KH, Barnewolt CE, Logvinenko T, Chow JS. Interobserver and Intra-Observer Reliability of the Urinary Tract Dilation Classification System in Neonates: A Multicenter Study. J Urol. 2019 Jun;201(6):1186-1192. doi: 10.1097/JU.0000000000000026. PMID 30676479
- [Background] Gray MC, Zillioux JM, Varda B, Herndon CDA, Kurtz MP, Chow JS, Kern NG. Assessment of urinary tract dilation grading amongst pediatric urologists. J Pediatr Urol. 2020 Aug;16(4):457.e1-457.e6. doi: 10.1016/j.jpurol.2020.04.025. Epub 2020 Apr 30. PMID 32430210
- [Background] Suson KD, Preece J. Do current scientific reports of hydronephrosis make the grade? J Pediatr Urol. 2020 Oct;16(5):597.e1-597.e6. doi: 10.1016/j.jpurol.2020.04.003. Epub 2020 Apr 10. PMID 32345558
- [Background] Maizels M, Braga L, Gong EM, Liu D, Meade P, Nelson LD, Dungan JS. "1 Voice": Learn urinary tract dilation (UTD) classification to assess fetal & newborn urological ultrasound findings. J Pediatr Urol. 2017 Dec;13(6):559-562. doi: 10.1016/j.jpurol.2017.11.002. No abstract available. PMID 29248273

DOCUMENTS (2):
  • Study Protocol (2023-12-19): https://cdn.clinicaltrials.gov/large-docs/23/NCT06317623/Prot_000.pdf
  • Informed Consent Form (2023-12-19): https://cdn.clinicaltrials.gov/large-docs/23/NCT06317623/ICF_001.pdf